CLINICAL TRIAL: NCT00471016
Title: An Intervention to Improve End of Life Decision Making Among Homeless Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 0210S34223
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2007-05-08 (Estimated); Status verified 2007-05

CONDITIONS: End of Life Decision Making; Advance Care Planning

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Guided intervention

SUMMARY:
This project is a prospective, randomized controlled trial to improve the end of life experience for homeless persons by facilitating the expression of their wishes and enhancement of their dignity when facing serious illness, death, or the prospect of dying. Our main hypothesis is that homeless persons will engage in this intervention and increase rates of advance directive completion.

DETAILED DESCRIPTION:
This project is a prospective, randomized controlled trial to improve the end of life experience for homeless persons by facilitating the expression of their wishes and enhancement of their dignity when facing serious illness, death, or the prospect of dying. Our main hypothesis is that homeless persons will engage in this intervention and increase rates of advance directive completion.

Participants were recruited from Listening House, a drop-in center for homeless individuals located in St. Paul, Minnesota and represent a convenience sample. Participants were required to speak English, not be overtly intoxicated, and have been homeless during the previous six months. The study was reviewed and approved by the institutional review board of the University of Minnesota. All participants who entered the study gave written and oral consent for randomization and data measurement and screening.

After recruitment and consent, participants were randomized into two intervention arms, minimal intervention (MI) and guided intervention (GI). All participants received educational materials about advance directives and advance care planning, pre-intervention surveys, and an advance care planning document, designated HELP, specifically designed for marginalized populations to preserve autonomy and elicit preferences of EOL care.

All participants completed a baseline written pre-test and survey. For this, they received compensation of $5. Those randomized to the minimal intervention were provided the opportunity to complete a HELP document if they so desired. Participants randomized to the GI group were provided with the written instructions and tools and asked to return to meet with investigators for one-on-one counseling and assistance in completion of the HELP document on one of several days later during the week of enrollment. Three months after enrollment, post-intervention evaluations were sought from both MI and GI subjects. There was no financial incentive offered for completion of the HELP form.

Measurement The primary outcome of interest was the completion of a legally valid advance directive, the HELP document, which was measured by inspection of HELP documents as well as self-report. Secondary outcomes include knowledge, attitude, and behavior variables measured through a questionnaire administered at baseline and at follow-up. Demographic information, including education and living situations, was also collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Homeless in last six months
* Speak English
* Age 18-65

Exclusion Criteria:

* Intoxicated
* Minor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2006-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Completion of an advance directive | Three months

SECONDARY OUTCOMES:
Knowledge, attitude, and behavioral measures | Three months

CONTACTS AND LOCATIONS:
Overall Officials: John Y Song, MD, Principal Investigator — University of Minnesota
Locations (1):
- Listening House, Saint Paul, Minnesota, United States